CLINICAL TRIAL: NCT05079477
Title: Communicating the Health Risks of Sugar-Sweetened Beverages: A Randomized-controlled Experiment of Different Nutrition Labels on Purchases and Consumption
Brief Title: Online Study of the Effects of Sugary Drink Warning Labels on Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 844786; R01DK111558 (NIH)
Record Dates: First submitted 2021-09-15; First posted 2021-10-15 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Food Preferences
Keywords: food labeling; child; sugar-sweetened beverages; eating; drinking; choice behavior
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Intervention Model Description: This randomized, controlled online study will capture beverage and snack purchases from an online store. These products will be mailed to participants for each of the 4 shopping weeks. Participants' consumption will be measured at the beginning and end of the study. As this is a within-participant study, consumption for each arm will be compared to baseline for that participant (Week 1 shopping).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calorie label (Active Comparator): Calorie label (control) will display a calories per package label on all beverages, not just sugary drinks. This is modeled after the American Beverage Association's current "Clear on Calories" labels. Additionally, all snack items will have a calories per serving label.
  Interventions: Behavioral: Exposure to calorie information
- Sugar graphic warning label (Experimental): All products in this arm will also have calorie labels. Beverages with added sugar will also have sugar graphic warning labels with the text: "WARNING: drinking beverages with added sugars contributes to obesity, diabetes, and tooth decay" along with graphics depicting the amount of sugar in the beverage.
  Interventions: Behavioral: Exposure to sugar-sweetened beverage warning labels; Behavioral: Exposure to calorie information

INTERVENTIONS:
Behavioral: Exposure to sugar-sweetened beverage warning labels — Graphic images of the amount of sugar (randomly assigned teaspoons, packets, or cubes) and text warning labels
  Arms: Sugar graphic warning label
Behavioral: Exposure to calorie information — Calories for all beverages and foods

SUMMARY:
The aim of this study is to determine the degree to which sugar-sweetened beverages (SSB) warning labels increase consumers' knowledge about the potential health harms of SSBs and reduce SSB purchases and consumption. 216 racially and ethnically diverse parents of children 6-11 years old will be recruited to buy snacks and beverages for four weeks via an online store that ships participants their purchases. Participants will be randomized to either 1) calorie labels (control); or 2) sugar graphic warning labels. The investigators hypothesize that sugar graphic warning labels displayed in an online store in weeks 2-4 will lead to the greatest reductions from week 1 across both primary outcomes compared to the control group that will only see calorie labels.

DETAILED DESCRIPTION:
During this study, participants will shop in an online store created using Shopify for four weeks. In this within-participant design, the first week of shopping is baseline. Participants will then be randomized to different store interfaces for the remaining three weeks based on one of two warning label conditions: 1) calorie labels (control); or 2) sugar graphic warning labels. Participants will complete a brief survey at the start of the study to assess demographic information, information about parent and child beverage consumption, and their online shopping experiences. At the end they will complete another survey about their beverage consumption, their experience shopping in the store, whether they noticed and used the warning labels, and their ability to recall the warning label message. Participants will also be asked about their perceptions of a specific type of warning label in this final survey. Upon completion of the survey, participants will be shown a debriefing statement explaining the study purpose. After they read the information, they will be asked whether or not they consent to allow their data to be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* a primary caregiver of a child 6-to-11 years old;
* >=18 years old;
* can read and speak English;
* primary grocery shopper for their household;
* have regular Internet access; and
* report that the oldest of their children between 6 and 11 years old is consuming sugar sweetened beverages at least twelve times per month or approximately three times a week

Exclusion Criteria:

* not a primary caregiver of a child 6-to-11 years old;
* <18 years old;
* cannot read and/or speak English;
* not the primary grocery shopper for their household;
* does not have regular Internet access; and
* does not report that the oldest of their children between 6 and 11 years old is consuming sugar sweetened beverages at least twelve times per month or approximately three times a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Roberto, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
In the consenting process, participants agreed that de-identified data produced from this project may be distributed for future research studies without additional informed consent. Any de-identified data shared will be done so via PennBox, a secure method to transfer files.
Supporting Information: SAP
Time Frame: starting 6 months after publication
Access Criteria: The PI will review requests to use de-identified study data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited online from October 2021 to November 2022.
Pre-assignment Details: Of the 216 participants, 2 were pilot participants who helped us discover some necessary changes to study procedures. They were excluded from analysis along with 2 lost to follow-up, 1 who withdrew, and 22 participants who were not confirmed eligible with baseline measures, leaving 189 participants for analysis.
Period: Overall Study
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Started | 108 | 108
Completed | 94 | 95
Not Completed | 14 | 13
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ineligible based on baseline survey (eligible based on protocol: recruitment screener) | 11 | 11
Not completed — Ineligible because pilot participants. The protocol changed after running them. | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calorie Label | Sugar Graphic Warning Label | Total
Number analyzed (Participants) | 108 | 108 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (7) | 40 (7) | 40 (7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 8 | 7 | 15
  Gender: Female | 97 | 101 | 198
  Gender: Non-binary / Gender non-conforming | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 101 | 105 | 206
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 48 | 86
  White | 57 | 53 | 110
  More than one race | 8 | 5 | 13
  Unknown or Not Reported | 2 | 1 | 3
Education level [Count of Participants; unit: Participants]
  Less than high school | 1 | 2 | 3
  High school graduate or received GED | 9 | 12 | 21
  Associates degree | 9 | 15 | 24
  Some college | 18 | 13 | 31
  College/University degree | 32 | 32 | 64
  Graduate or professional education | 39 | 34 | 73
Number of children in household [Count of Participants; unit: Participants]
  1 child | 29 | 15 | 44
  2 children | 48 | 50 | 98
  3 children | 17 | 26 | 43
  4 or more children | 14 | 17 | 31
Number of adults in household [Count of Participants; unit: Participants]
  1 adult | 32 | 32 | 64
  2 adults | 61 | 62 | 123
  3 or more adults | 15 | 14 | 29
Marital status [Count of Participants; unit: Participants]
  Married or living with partner | 73 | 64 | 137
  Single (never married, divorced, widowed, separated) | 35 | 44 | 79

OUTCOME MEASURES:

1. Primary Outcome: Beverage Calories Purchased, Week 1
Description: Logged beverage calories/100mL purchased. Number of servings per item and number of items per package varied by product; therefore, calorie amounts were standardized to calories/100mL for beverages.
Time Frame: one week
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener). 3 participants did not have order data because did not shop any of the 4 weeks.
Measure: Mean (Standard Deviation); unit: Logged calories/100mL
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Logged calories/100mL | 1.43 (0.62) | 1.40 (0.62)

2. Primary Outcome: Beverage Calories Purchased, Weeks 2-4
Description: Logged average beverage calories/100mL purchased per week over Weeks 2-4. Number of servings per item and number of items per package varied by product; therefore, calorie amounts were standardized to calories/100mL for beverages.
Time Frame: three weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Logged calories/100mL
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Logged calories/100mL | 1.49 (0.50) | 1.43 (0.48)

3. Primary Outcome: Beverage Added Sugars Purchased, Week 1
Description: Beverage grams of added sugars/100mL purchased. Number of servings per item and number of items per package varied by product; therefore, added sugar amounts were standardized to grams of added sugar/100mL for beverages.
Time Frame: one week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/100mL
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
g/100mL | 8.95 (8.75) | 8.10 (8.43)

4. Primary Outcome: Beverage Added Sugars Purchased, Weeks 2-4
Description: Average beverage grams of added sugars/100mL purchased per week over Weeks 2-4. Number of servings per item and number of items per package varied by product; therefore, added sugar amounts were standardized to grams of added sugar/100mL for beverages.
Time Frame: three weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/100mL
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
g/100mL | 8.90 (8.07) | 6.99 (7.06)

5. Secondary Outcome: Number Purchasing a Sweetened Beverage, Week 1
Description: Number of parents buying a sweetened beverage within each condition
Time Frame: one week
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Participants | 67 | 68

6. Secondary Outcome: Number Purchasing a Sweetened Beverage, Weeks 2-4
Description: Number of parents buying a sweetened beverage at any point during Weeks 2-4, within each condition
Time Frame: three weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Participants | 77 | 73

7. Secondary Outcome: Snack Calories Purchased, Week 1
Description: Logged snack calories/100g purchased. Number of servings per item and number of items per package varied by product; therefore, calorie amounts were standardized to calories/100g for snacks.
Time Frame: one week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Logged calories/100g
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Logged calories/100g | 2.89 (0.22) | 2.94 (0.22)

8. Secondary Outcome: Snack Calories Purchased, Weeks 2-4
Description: Logged average snack calories/100g purchased per week over Weeks 2-4. Number of servings per item and number of items per package varied by product; therefore, calorie amounts were standardized to calories/100g for snacks.
Time Frame: three weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Logged calories/100g
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Logged calories/100g | 2.94 (0.21) | 2.96 (0.20)

9. Secondary Outcome: Snack Added Sugars Purchased, Week 1
Description: Snack grams of added sugars/100g purchased. Number of servings per item and number of items per package varied by product; therefore, added sugar amounts were standardized to grams of added sugar/100g for snacks.
Time Frame: one week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/100g
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
g/100g | 28.3 (28.0) | 31.2 (29.0)

10. Secondary Outcome: Snack Added Sugars Purchased, Weeks 2-4
Description: Average snack grams of added sugars/100g purchased per week over Weeks 2-4. Number of servings per item and number of items per package varied by product; therefore, added sugar amounts were standardized to grams of added sugar/100g for snacks.
Time Frame: three weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/100g
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
g/100g | 38.3 (32.1) | 37.3 (26.0)

11. Secondary Outcome: Total Calories Purchased, Week 1
Description: Log of the summed beverage and snack calories purchased
Time Frame: one week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Logged calories
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Logged calories | 3.52 (0.26) | 3.55 (0.22)

12. Secondary Outcome: Total Calories Purchased, Weeks 2-4
Description: Log of the average summed beverage and snack calories purchased per week over Weeks 2-4
Time Frame: three weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Logged calories
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Logged calories | 3.56 (0.22) | 3.55 (0.22)

13. Secondary Outcome: Total Added Sugars Purchased, Week 1
Description: Summed grams of beverage and snack added sugars purchased
Time Frame: one week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Grams | 353 (300) | 321 (260)

14. Secondary Outcome: Total Added Sugars Purchased, Weeks 2-4
Description: Average summed grams of beverage and snack added sugars purchased per week over Weeks 2-4
Time Frame: three weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Grams | 378 (277) | 327 (238)

15. Secondary Outcome: Volume of Sweetened Beverages Consumed by Child, Baseline
Description: Ounces of sweetened beverages (labeled in sugar condition) consumed per day in the last month by the child as measured by the Beverage Intake Questionnaire (BEV-Q) parent self-report survey.
Time Frame: baseline
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener).
Measure: Median (Full Range); unit: Ounces
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 97 | 95
Ounces | 6.4 [0 to 192] | 7.2 [0 to 240]

16. Secondary Outcome: Volume of Sweetened Beverages Consumed by Child, Final
Description: as for outcome 15
Time Frame: Week 4
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener). 3 participants did not have final survey data.
Measure: Median (Full Range); unit: Ounces
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Ounces | 6.4 [0 to 156] | 7.2 [0 to 240]

17. Secondary Outcome: Volume of Sweetened Beverages Consumed by Parent, Baseline
Description: Ounces of sweetened beverages (labeled in sugar condition) consumed per day in the last month by the parent as measured by the Beverage Intake Questionnaire (BEV-Q) self-report survey.
Time Frame: baseline
Population: as for outcome 15
Measure: Median (Full Range); unit: Ounces
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 97 | 95
Ounces | 4 [0 to 200] | 6 [0 to 240]

18. Secondary Outcome: Volume of Sweetened Beverages Consumed by Parent, Final
Description: as for outcome 17
Time Frame: Week 4
Population: as for outcome 16
Measure: Median (Full Range); unit: Ounces
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 95
Ounces | 3.4 [0 to 160] | 5.6 [0 to 240]

19. Secondary Outcome: Noticing the Label
Description: Participants will respond "yes," "no," or "I don't know" to the item: "When you selected a beverage to purchase in the store, did you notice any labels on the beverages other than calorie information?"
Time Frame: Week 4
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener). 3 participants did not have final survey data, and 1 person didn't answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 94
Participants
  Yes | 34 | 62
  No | 48 | 22
  Don't know | 12 | 10

20. Secondary Outcome: Perceived Label Influence
Description: Participants will respond: "yes", "no," or "I did not notice any labels" in response to the question of whether the label influenced their purchase.
Time Frame: Week 4
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener). 3 participants did not have final survey data. And 1 person didn't answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 94
Participants
  Yes | 15 | 41
  No | 19 | 21
  I did not notice any labels | 60 | 32

21. Secondary Outcome: How Much do You Trust the Information on This Label
Description: "How much do you trust the information on this label?". Responses will be measured with a 7-point Likert scale where 1=Not at all and 7=Extremely. Higher numbers indicate greater trust in the label.
Time Frame: Week 4
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener). 3 participants did not have final survey data. And 3 more who didn't answer this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 93
units on a scale | 5.4 (1.7) | 6.0 (1.3)

22. Secondary Outcome: Likelihood of Label Changing Thoughts
Description: "If this government warning label were on a beverage, how much would it change your thoughts about the healthiness of that beverage for your child?" Responses will be measured with a 5-point Likert scale where 1=Not at all and 5=A lot. Higher numbers indicate the label would be more likely to change perceptions of beverage healthiness.
Time Frame: Week 4
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener). 3 participants did not have final survey data. Three more didn't answer this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 93
units on a scale | 3.7 (1.4) | 4.2 (1.0)

23. Secondary Outcome: Encourage You to Give Fewer Beverages to Your Child
Description: "If you saw this government warning label on a beverage, would the label encourage you to serve your child that beverage less often?" Responses will be measured with a 5-point Likert scale where 1=Definitely no and 5=Definitely yes. Higher numbers indicate greater likelihood of serving unhealthy beverages less often.
Time Frame: Week 4
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener). 3 participants did not have final survey data. 3 additional didn't answer this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 93
units on a scale | 3.9 (1.2) | 4.3 (1.1)

24. Secondary Outcome: Negative Reactions to the Label
Description: Average negative emotional response to the label will be examined (said the warning label made them feel worried, fearful, guilty, or disgusted or grossed out). Responses will be measured with a 5-point Likert scale averaging across the 4 negative emotions where 1=Not at all and 5=Extremely. Higher numbers indicate more negative reactions.
Time Frame: Week 4
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener). 3 participants did not have final survey data. Three additional participants didn't answer this question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 93
score on a scale | 2.4 (0.9) | 3.4 (0.9)

25. Secondary Outcome: Child Enjoyment of Water
Description: "How much do you think your child would enjoy this product?" Responses will be measured with a 7-point Likert scale where 1=Not at all and 7=Extremely. Higher numbers indicate greater enjoyment of the product.
Time Frame: Week 4
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener). 3 participants did not have final survey data. And participants who did not answer this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 94
units on a scale | 5.1 (1.9) | 5.2 (2.0)

26. Secondary Outcome: Child Enjoyment of Orange Juice
Description: as for outcome 25
Time Frame: Week 4
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
units on a scale | 5.3 (1.8) | 5.1 (1.8)

27. Secondary Outcome: Child Enjoyment of Soda
Description: as for outcome 25
Time Frame: Week 4
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
units on a scale | 4.8 (2.5) | 4.4 (2.5)

28. Secondary Outcome: Child Enjoyment of Sports Drink
Description: as for outcome 25
Time Frame: Week 4
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 93
units on a scale | 4.6 (2.1) | 4.7 (2.3)

29. Secondary Outcome: Likely to Serve or Buy Water
Description: "How likely are you to serve or buy this product for your child in the next 4 weeks?" Responses will be measured with a 7-point Likert scale where 1=Not at all and 7=Extremely. Higher numbers indicate greater likelihood of serving or buying the product for their child.
Time Frame: Week 4
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 94 | 94
units on a scale | 4.0 (2.4) | 4.0 (2.5)

30. Secondary Outcome: Likely to Serve or Buy Orange Juice
Description: as for outcome 29
Time Frame: Week 4
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
units on a scale | 4.1 (2.1) | 4.1 (2.1)

31. Secondary Outcome: Likely to Serve or Buy Soda
Description: as for outcome 29
Time Frame: Week 4
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
units on a scale | 2.1 (1.6) | 2.1 (1.7)

32. Secondary Outcome: Likely to Serve or Buy Sports Drinks
Description: as for outcome 29
Time Frame: Week 4
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 93
units on a scale | 2.6 (1.9) | 2.8 (1.8)

33. Secondary Outcome: Health Beliefs and Risk Perceptions Index for Water
Description: Summed responses to the following 7 health perception questions, 6 of which are prompted with the statement "Drinking this product often would…". The statements end with the following health belief and risk perception language: "lead my child to gain weight," "increase my child's risk of heart disease," "increase my child's risk of diabetes," "make my child feel energized," "help my child focus at school", and "help my child live a healthy life." The other item is: "How healthy do you think this product is for your child?" Responses to questions about weight gain, heart disease, and diabetes will be reverse coded, so higher scores on the summed index will indicate a stronger positive health perception of the beverages. This index ranges 7 to 49.
Time Frame: Week 4
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener). 3 participants did not have final survey data. And participants who did not answer these questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
score on a scale | 41.8 (5.7) | 40.3 (6.7)

34. Secondary Outcome: Health Beliefs and Risk Perceptions Index for Orange Juice
Description: as for outcome 33
Time Frame: Week 4
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
score on a scale | 28.7 (7.9) | 29.3 (7.4)

35. Secondary Outcome: Health Beliefs and Risk Perceptions Index for Soda
Description: as for outcome 33
Time Frame: Week 4
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
score on a scale | 13.4 (5.4) | 14.6 (5.9)

36. Secondary Outcome: Health Beliefs and Risk Perceptions Index for Sports Drinks
Description: as for outcome 33
Time Frame: Week 4
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 93
score on a scale | 23.3 (6.8) | 23.1 (7.1)

37. Secondary Outcome: Estimate of How Many Teaspoons of Added Sugar Are in Water
Description: This variable will be measured continuously based on a text box provided to participants. Median teaspoons in each condition will be assessed
Time Frame: Week 4
Population: Excludes 22 participants who were not eligible according to the baseline survey (although met protocol eligibility with recruitment screener). 3 participants did not have final survey data. Additional participants who did not answer this question.
Measure: Median (Full Range); unit: teaspoons
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
teaspoons | 0 [0 to 10] | 0 [0 to 32]

38. Secondary Outcome: Estimate of How Many Teaspoons of Added Sugar Are in Orange Juice
Description: as for outcome 37
Time Frame: Week 4
Population: as for outcome 37
Measure: Median (Full Range); unit: teaspoons
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
teaspoons | 4 [0 to 120] | 4 [0 to 60]

39. Secondary Outcome: Estimate of How Many Teaspoons of Added Sugar Are in Soda
Description: as for outcome 37
Time Frame: Week 4
Population: as for outcome 37
Measure: Median (Full Range); unit: teaspoons
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
teaspoons | 10 [2 to 200] | 16 [0 to 120]

40. Secondary Outcome: Estimate of How Many Teaspoons of Added Sugar Are in Sports Drinks
Description: as for outcome 37
Time Frame: Week 4
Population: as for outcome 37
Measure: Median (Full Range); unit: teaspoons
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 93
teaspoons | 6 [0 to 60] | 8 [0 to 30]

41. Secondary Outcome: Perceived Amount of Added Sugar in Water
Description: This variable will be measured with a 3-point ordinal Likert scale with values: 1 = "too little for my child", 2 = "just right for my child" and 3 = "too much for my child". Higher scores indicate beverage is perceived as having too much added sugar.
Time Frame: Week 4
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
units on a scale | 2.0 (0.4) | 2.1 (0.4)

42. Secondary Outcome: Perceived Amount of Added Sugar in Orange Juice
Description: as for outcome 41
Time Frame: Week 4
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
units on a scale | 2.5 (0.5) | 2.4 (0.5)

43. Secondary Outcome: Perceived Amount of Added Sugar in Soda
Description: as for outcome 41
Time Frame: Week 4
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 94
units on a scale | 3.0 (0.3) | 3.0 (0.2)

44. Secondary Outcome: Perceived Amount of Added Sugar in Sports Drinks
Description: as for outcome 41
Time Frame: Week 4
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calorie Label | Sugar Graphic Warning Label
Number analyzed (Participants) | 93 | 93
units on a scale | 2.7 (0.5) | 2.7 (0.5)

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Calorie Label | Sugar Graphic Warning Label
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/108
Other Adverse Events (participants affected / at risk) | 0/108 | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT05079477/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT05079477/ICF_000.pdf